CLINICAL TRIAL: NCT04612907
Title: A Randomized Phase III, Multicenter Study to Evaluate Different Fractionation Schedules of Radiotherapy to the Primary Tumour in Metastatic Hormone Sensitive Prostate Cancer
Brief Title: Different Fractionation Schedules of Radiotherapy to the Primary Tumour in Metastatic Hormone Sensitive Prostate Cancer
Acronym: Hypo-M1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hypo-M1 1.0
Record Dates: First submitted 2020-10-20; First posted 2020-11-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer; Radiotherapy Side Effect; Metastatic Cancer
Keywords: Metastatic prostate cancer radiotherapy primary tumor
MeSH Terms: conditions — Prostatic Neoplasms; Radiation Injuries; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to one of two treatment fractionations of radiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate hypo-fractionation (Active Comparator): Radiotherapy to the prostate delivered in 3Gy fractions x 19
  Interventions: Radiation: Moderate hypo-fractionation
- Ultra hypo-fractionation (Experimental): Radiotherapy to the prostate delivered in 6.1Gy fractions x 6
  Interventions: Radiation: Ultra-hypo-fractionation

INTERVENTIONS:
Radiation: Moderate hypo-fractionation — Patients will receive four weeks of radiotherapy
  Arms: Moderate hypo-fractionation
Radiation: Ultra-hypo-fractionation — Patients will receive two and a half weeks of radiotherapy
  Arms: Ultra hypo-fractionation

SUMMARY:
de Novo metastatic prostate cancer with limited metastatic spread benefits from local radiotherapy to the prostate. Two different fractionation schedules will be tested.

DETAILED DESCRIPTION:
Patients with de Novo metastatic prostate cancer with limited disease spread has been shown to gain benefit from local radiotherapy to the prostate. The internationally accepted fractionation schedule is 3 Gy (Gray) x 19-20 over a course of 4 weeks.

There is continous evidence for even more hypo-fractionated radiotherapy with higher fractionation doses. We will test if the schedule of 6.1Gy x 6 compares to standard of 3 Gy x 19 with regard to patient reported side-effects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Histological confirmed prostate cancer
3. Indication for early palliative radiation therapy of low burden metastatic prostate cancer. Low burden as defined by modified CHAARTED trial criteria to maximum 4 skeletal mets at any site and/or any number of lymph nodes
4. baseline E-PROM

Exclusion Criteria:

1. High burden metastatic prostate cancer including all with visceral mets.
2. Unable to comply with study procedures.
3. Other diseases or medication that will put the patient at risk for more toxicity from radiotherapy
4. Radiation treatment start later than nine months after the prostate cancer diagnosis.
5. Severe micturition problems, IPSS > 20 ( International Prostate Symptom Score)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer is a male disease
Enrollment: 420 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Toxicity as scored by PROM (Patient Reported Outcome Measures) at 8 weeks | 8 weeks
  Acute toxicity score by PROM at eight weeks post radiotherapy. The mean PCSS (Prostate Cancer Symptom Scale) bother score for urinary tract will be measured. The primary outcome measurement will be the difference between mean values in the respective treatment arms measured at 8 weeks after end of radiotherapy
Toxicity as scored by PROM at 8 weeks | 8 weeks
  Acute toxicity score by PROM at eight weeks post radiotherapy. The mean PCSS bother score for bowel will be measured. The primary outcome measurement will be the difference between mean values in the respective treatment arms measured at 8 weeks after end of radiotherapy

SECONDARY OUTCOMES:
Failure free survival | 12 months, 36 months
  To evaluate the proportion of patients that are failure free at 12 and 36 months, failure free survival (FFS)

CONTACTS AND LOCATIONS:
Overall Officials: Camilla of T Karlsson, Principal Investigator — Cancercentrum Umeå University
Locations (1):
- Cancercenter University hospital of Umeå, Umeå, Sweden